CLINICAL TRIAL: NCT02240615
Title: The Sinopsys Lacrimal Stent Used During the Repair of the Lacrimal System in Patients With Epiphora
Brief Title: The Sinopsys Lacrimal Stent for Lacrimal System Repair in Epiphora
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sinopsys Surgical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SLS-US-01
Record Dates: First submitted 2014-09-11; First posted 2014-09-15 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Epiphora
Keywords: Epiphora; Lacrimal Stent; Lacrimal System
MeSH Terms: conditions — Lacrimal Apparatus Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sinopsys Lacrimal Stent (Experimental): All enrolled patients will receive a Sinopsys Lacrimal Stent inserted from the caruncle to the ethmoid sinus. Discharge instructions will include administration of sterile saline and ophthalmic drops as well as assessments for device patency.
  Interventions: Device: Sinopsys Lacrimal Stent

INTERVENTIONS:
Device: Sinopsys Lacrimal Stent — Procedural insertion of the Sinopsys Lacrimal Stent in patients with epiphora

SUMMARY:
Prospective, open label, multi-center, non-randomized study designed to collect initial clinical data related to the safety and clinical performance of the Sinopsys Lacrimal Stent for use during repair of the lacrimal system in patients with functional or obstructive epiphora.

DETAILED DESCRIPTION:
Up to 10 patients will be enrolled and followed for six months. The primary objective is to demonstrate the safety and clinical performance of the Sinopsys Lacrimal Stent for use during repair of the lacrimal system for ethmoid sinus intubation and bypass to canalicular pathologies in this patient population. The primary outcome measure for performance is the relief of epiphora determined by both investigator assessment of stent patency and patient self-assessment of epiphora symptom improvement compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

* Clinically significant functional epiphora for at least three months
* Keros classification 1 or 2 skull base anatomy

Exclusion Criteria:

* Active infection
* Craniofacial deformity
* Severe inflammatory disease

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-10; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Relief of epiphora, determined by both 1) the Investigator assessment of the patency/function of the Sinopsys Lacrimal Stent ( and 2) the subject's self-assessment of tearing. | Six Months
  PI self assessment of stent patency and patient self assessment of improvement of epiphora symptoms compared to baseline

SECONDARY OUTCOMES:
Measurement of device insertion success | Procedural
Evaluation of all safety | Six Months
  Recording of all safety events that occur in the first six months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Harry Ross, MD, Study Director — Sinopsys Surgical Inc.; Teena Augostino, Study Director — Sinopsys Surgical Inc.
Locations (4):
- United States (4):
  - Stanford University, Stanford, California
  - University of Colorado Health Sciences Center, Aurora, Colorado
  - Center for Sight, Sarasota, Florida
  - Eye Care Specialists, Kingston, Pennsylvania